CLINICAL TRIAL: NCT05145348
Title: Prospective Monitoring of Antibody Response Following COVID-19 Vaccination in Patients With Down Syndrome
Acronym: PRIDE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: UMC Utrecht (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); National Institute for Public Health and the Environment (RIVM) (Other Government); Stichting Downsyndroom (SDS) (Unknown); Sanquin Research & Blood Bank Divisions (Other)
Responsible Party: Principal Investigator, Louis Bont, Clinical Professor, Principal investigator, UMC Utrecht
Other Study IDs: NL76336.041.21
Record Dates: First submitted 2021-12-03; First posted 2021-12-06 (Actual); Last update posted 2021-12-30 (Actual); Status verified 2021-12

CONDITIONS: Down Syndrome; SARS-CoV-2 Vaccination
Keywords: Down Syndrome; SARS-CoV-2 vaccination; Immuneresponse
MeSH Terms: conditions — Down Syndrome | interventions — BNT162 Vaccine; ChAdOx1 nCoV-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, Whole blood, PBMC's, mucosal nose swab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Down syndrome, adults: Adults and adolescents with Down syndrome >16 years old.
  Interventions: Biological: Immune response to Sars-CoV-2 vaccinations; including COVID-19 vaccin Moderna, Comirnaty (Pfizer) and Vaxzevria (AstraZeneca)
- Healthy control, adults: Healthy adults and adolescents without Down syndrome > 16 years old. Without any significant comorbidities.
  Interventions: Biological: Immune response to Sars-CoV-2 vaccinations; including COVID-19 vaccin Moderna, Comirnaty (Pfizer) and Vaxzevria (AstraZeneca)
- Down syndrome, children: Children with Down syndrome < 16 years old.
  Interventions: Biological: Immune response to Sars-CoV-2 vaccinations; including COVID-19 vaccin Moderna, Comirnaty (Pfizer) and Vaxzevria (AstraZeneca)
- Healthy control, children: Healthy children without Down syndrome < 16 years old. Without any significant comorbidities.
  Interventions: Biological: Immune response to Sars-CoV-2 vaccinations; including COVID-19 vaccin Moderna, Comirnaty (Pfizer) and Vaxzevria (AstraZeneca)

INTERVENTIONS:
Biological: Immune response to Sars-CoV-2 vaccinations; including COVID-19 vaccin Moderna, Comirnaty (Pfizer) and Vaxzevria (AstraZeneca) — The vaccination is not part of the study, but part of the national immunization programme of the Netherlands. Blood will be drawn at 4 time points: baseline (t=1, <2 months prior to first vaccination); t=2: 21-28 days after first vaccination and prior to second vaccination; t=3: 28 (21-42) days after second vaccination; t=4: 12 months (+/- 1 month) after second vaccination. Mucosal Lining Fluid (MLF) samples will be collected at 28 days (3-6 weeks) (t=3) and 12 (+/- 1) months (t=4) after the second vaccination.

SUMMARY:
The risk of severe course of SARS-CoV-2 infection in people with Down Syndrome is substantially increased. The risk of death is 3-10 fold higher than in healthy people. SARS-CoV-2 vaccines have been registered for adults and adolescents but none of them have been studied in people with Down Syndrome. Vaccine responses in people with Down Syndrome are known to be suboptimal. Therefor the objective of this study is to assess the immunogenicity of SARS-CoV-2 vaccination in people with Down syndrome.

To do so, the antibody response, cellulair and mucosal immuneresponse in people with Down syndrome after the SARS-CoV-2 vaccination will be evaluated and compared to healthy controls.

DETAILED DESCRIPTION:
All participants will receive two vaccinations against COVID-19 according to the manufacturer's instructions as part of the Dutch SARS-CoV-2 vaccination program (GGD/RIVM). To assess the immune response after vaccination, blood samples will be collected at baseline (i.e. <2 months prior to first vaccination (t=1)), 21-28 days after first vaccination and prior to second vaccination (t=2), 28 days (3-6 weeks) (t=3) and 12 (+/- 1) months (t=4) after the second vaccination. To evaluate haematological parameters, additional blood samples will be collected at baseline, 21-28 days after the first vaccination and 28 days after the second vaccination. Per visit/time-point maximum 60 ml blood will be drawn. In children the maximum amount of blood taken per visit/time-point will be 0,8 ml/kg up to 60 ml. In addition Mucosal Lining Fluid (MLF) samples will be collected at 28 days (3-6 weeks) (t=3) and 12 (+/- 1) months (t=4) after the second vaccination to evaluate the mucosal immune response after SARS-CoV-2 vaccination. In the pediatric part of the study Mucosal Lining Fluid (MLF) samples will be collected at all timepoints.

Although vaccine administration is not part of this study, vaccine type, batch number and dosing will be registered. This information will be obtained from the "COVID-vaccination information and monitoring system (CIMS)" of the RIVM.

Clinical course including the occurrence of COVID-19 will be monitored during the first year after vaccination. To evaluate vaccination related AEs, patients will be asked to collect solicited local and systemic AEs for 7 days after each vaccination using an online questionnaire, as vaccination related AEs are mainly expected in the first week after vaccination. The link to the online questionnaires will be sent to the emailaddress of the participants and/or their representative/carer. If the participants and/or their representative/carers are not able to fill out the diary online, they will be contacted by phone.

Although this study is not powered to detect differences in protection against COVID-19 between patients and controls, information on incidence of SARS-CoV-2 infection, outcome of COVID-19 will be collected up to 12 months after vaccination for descriptive purposes.

ELIGIBILITY:
Inclusion Criteria:

* Willing to receive routine COVID-19 vaccination with Pfizer, Moderna or AstraZeneca vaccine.
* Age: ≥12 years or < 12 years once vaccine is recommended for routine use in the respective age group
* Either Down syndrome (DS) or household contacts without DS of participant with DS.

Exclusion Criteria:

Down syndrome cohort:

* History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (e.g. anaphylaxis) to any component of the study intervention(s).
* Organ transplant recipients
* Active malignancy or completion of treatment for malignancy in previous 3 months
* Infection with Human Immunodeficiency Virus (HIV)
* Bleeding diathesis or condition associated with prolonged bleeding that would, in the opinion of the investigator, contraindicate intramuscular injection.

Healthy control cohort:

- As in Down Syndrome cohort

Plus:

* Active medical care for inherited or acquired immune deficiency
* Any severe comorbidity for which regular medical care is needed (e.g. heart failure, COPD, diabetes)

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Down syndrome:
  The patient population will either live in institutions or outside these facilitys depending on the cognitive functions and additional care needed. Children will mostly live with their parents. All participants will live in the Netherlands
  Healthy control:
  All healthy control participants will live in the Netherlands, no specific region.
Sampling Method: Probability Sample
Enrollment: 640 (Estimated)
Dates: Start 2021-02-03 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Antibody based immune response to vaccination against COVID-19 28 days (t=3) after the second vaccination as compared to controls. | 28 days after the second vaccination
  Participants will be classified as responders or non-responders. The definition of response will be based on the latest available data from the pivotal studies and will be defined prior to data analyses and the first database lock. The percentage of responders in the DS cohort will be compared with the percentage responders in the HS cohort.

SECONDARY OUTCOMES:
Longevity of SARS-CoV-2 specific antibodies | 1 year after the second vaccination
  Longevity of SARS-CoV-2 specific antibodies after the second vaccination will be compared between cohorts.
SARS-CoV2 specific T cell response | Number of T cells will be measured at baseline, at 21-28 days after the first vaccination and at 28 days after the second vaccination
  The number of IFN-ɣ producing SARS-CoV2 specific T cells/million PBMC (mean of 3 measures)
Mucosal SARS-CoV-2 specific antibodies | Mucosal antibodies will be measured 28 days and 12 months after the second vaccination.
  Antibody titers will be compared between cohorts and with antibody titers in blood

OTHER OUTCOMES:
Determination of fucosylation, sialylation, galactosylation and bisection of IgG in patients with a history of COVID-19. | All time points
  Determination of levels of fucosylation, sialylation, galactosylation and bisection of both bulk IgG and anti-SARS-CoV-2 S protein IgG in participants with a history of proven mild or severe COVID-19.
Age-specific T-cell immunophenotyping | All time points
  Immunophenotyping, in particular naïve T-cell counts will be measured.
Neutralizing capacity of SARS-CoV-2 antibodies | Measurements at baseline, 21-28 days after first vaccination and 28 days, and 12 months after second vaccination.
  Comparison of the neutralizing capacity of SARS-CoV-2 antibodies between cohorts
Incidence and outcome of SARS-CoV-2 infection | During time period of 12 months after vaccination.
  Incidence and outcome during period of 12 months after vaccination. For participants with a positive test, information about disease severity will be presented including hospital admissions, use of oxygen, intensive care admission and mechanical ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Louis J Bont, MD, PhD, Principal Investigator — UMC Utrecht
Locations (1):
- UMC utrecht, Utrecht, Netherlands

REFERENCES:
- [Derived] Streng BMM, Hensen LCM, Delemarre EM, Binnendijk RS, Smits G, den Hartog G, van der Klis FR, de Vries E, Burger JA, van Gils MJ, Coppus AMW, Weijerman ME, Lamberts R, de Graaf G, Bont LJ, Wildenbeest JG. Antibody concentration and function following SARS-CoV-2 vaccination decrease with age in adults and children with Down syndrome. Vaccine. 2026 Feb 15;73:128079. doi: 10.1016/j.vaccine.2025.128079. Epub 2025 Dec 24. PMID 41447779
- [Derived] Hensen LCM, Streng BMM, van Wijk F, Nierkens S, van Binnendijk RS, Buisman AM, Coppus AMW, Geurts van Kessel CH, de Graaf G, van der Klis FR, Lamberts R, Vidarsson G, Ruckwardt TJ, de Vries E, de Vries RD, Weijerman ME, Weinberger DM, Wildenbeest JG, Bont LJ, Delemarre EM. T-cell responses to SARS-CoV-2 vaccinations in adults with Down syndrome - a prospective cohort study. Hum Vaccin Immunother. 2025 Dec;21(1):2583416. doi: 10.1080/21645515.2025.2583416. Epub 2025 Nov 6. PMID 41196011
- [Derived] Streng BMM, Bont M, Delemarre EM, Binnendijk RS, Smit G, den Hartog G, Coppus AMW, de Vries E, Weijerman ME, Lamberts R, de Graaf G, van der Klis FR, Vidarsson G, Rave N, Bont LJ, Wildenbeest JG. Decreased Antibody Response After Severe Acute Respiratory Syndrome Coronavirus 2 Vaccination in Patients With Down Syndrome. J Infect Dis. 2022 Sep 4;226(4):673-677. doi: 10.1093/infdis/jiac235. PMID 35748853